CLINICAL TRIAL: NCT04353531
Title: An Observational Study to Investigate the Aerosol Particle Distribution During Aerosol Generating Procedures
Brief Title: Investigate the Aerosol Particle Distribution During Aerosol Generating Procedures
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: COVID19-aerosol
Record Dates: First submitted 2020-03-23; First posted 2020-04-20 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Transmission, Patient Professional; High-flow Nasal Cannula
MeSH Terms: interventions — Intubation; Tracheostomy; Respiratory Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: High-flow nasal cannula — High-flow nasal cannula is a modality of oxygen device that can provide gas flow meets or exceeds patient inspiratory flow demand (flow can be set at 10-60 L/min), it has been proven to improve oxygenation and reduce intubation rate in hypoxemic patients.
  Other Names: HFNC, high-flow high humidity nasal cannula
Device: Surgical mask — A procedure mask will be used to cover patient's face after HFNC is initiated.
  Other Names: procedure mask
Procedure: bronchoscopy examination — is a procedure that allows a doctor to examine the inside of the lungs, including the bronchi, which are the main pathways into the lungs. During a bronchoscopy, a doctor inserts a thin tube containing a light and camera into the lungs through the nose or mouth or via artificial airway such as intubation or tracheotomy tube
Procedure: intubation — Intubation is the process of inserting a tube, called an endotracheal tube (ET), through the mouth and then into the airway. This is done so that a patient can be placed on a ventilator to assist with breathing during anesthesia, sedation, or severe illness.
Procedure: tracheostomy — A tracheostomy is a medical procedure - either temporary or permanent - that involves creating an opening in the neck in order to place a tube into a person's windpipe. The tube is inserted through a cut in the neck below the vocal cords. This allows air to enter the lungs.
Device: nebulization — A nebulizer is a piece of medical equipment that a person with asthma or another respiratory condition can use to administer medication directly and quickly to the lungs
Diagnostic Test: Pulmonary function test — Pulmonary function tests (PFTs) are noninvasive tests that show how well the lungs are working. The tests measure lung volume, capacity, rates of flow, and gas exchange.

SUMMARY:
Massive number of clinicians were infected during the outbreak of COVID-19, which raised the concerns of utilizing "aerosol generating procedures", particularly the use of high-flow nasal cannula, noninvasive ventilation, intubation, bronchoscopy examination and pulmonary function test. There appears to be a trend to avoid those treatments. Instead, aggressive intubation might cause shortage of medical devices and add extra workload. Therefore, we aimed to do a clinical observational study to evaluate the aerosol generation in these procedures and explore the potential measures to reduce the aerosol generation or dispersion.

DETAILED DESCRIPTION:
The intent is to monitor exhaled aerosol produced by COVID-19 patients pre and post aerosol generating procedures. Monitoring will occur at a distance of 1 and 3 feet from the subject's airway. This observational study will be conducted in standard patient hospital rooms (standard or negative pressure room).

ELIGIBILITY:
Inclusion Criteria:

• Adult patients who are diagnosed as COVID-19 infection in ICU or Adult patients are indicated for pulmonary function tests

Exclusion Criteria:

• No need for any respiratory therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who are diagnosed as COVID-19 infection and admitted to adult ICU will be enrolled in Rush University Medical Center, Chicago, IL, USA. Patients will be excluded if patients do not require any respiratory treatments.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
The aerosol mass/count concentration pre procedure/treatment at 1 foot away from patient | 5 minutes before procedure/treatment
  The aerosol mass/count concentration pre procedure/treatment at 1 foot away from patient's airway in the patient's room
The virus load in the air sample pre procedure/treatment at 1 foot away from patient | 1 hour before procedure/treatment
  The virus load in the air sample pre procedure/treatment at 1 foot away from patient's airway in the patient's room
The virus load in the air sample during/after procedure/treatment at 1 foot away from patient | 1 hour during/after procedure/treatment
  The virus load in the air sample during/after procedure/treatment at 1 foot away from patient's airway in the patient's room
The aerosol mass/count concentration pre procedure/treatment at 3 feet away from patient | 5 minutes before procedure/treatment
  The aerosol mass/count concentration pre procedure/treatment at 3 feet away from patient's airway in the patient's room
The aerosol mass/count concentration and virus load in the air sample during procedure/treatment at 1 foot away from patient | during procedure/treatment
  The aerosol mass/count concentration and virus load in the air sample during procedure/treatment at 1 foot away from patient's airway in the patient's room
The aerosol mass/count concentration during procedure/ treatment at 3 feet away from patient | during procedure/treatment
  The aerosol mass/count concentration during procedure/ treatment at 3 feet away from HFNC in the patient's room
The aerosol mass/count concentration post procedure/ treatment at 1 foot away from patient | 5 minutes post procedure/treatment
  The aerosol mass/count concentration post procedure/ treatment at 1 foot away from HFNC in the patient's room
The aerosol mass/count concentration 5 mins post procedure/ treatment at 3 feet away from patient | 5 minutes post procedure/treatment
  The aerosol mass/count concentration 5 mins procedure/ treatment at 3 feet away from HFNC in the patient's room

CONTACTS AND LOCATIONS:
Overall Officials: Jie Li, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush university medical center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data may be shared for research purpose based on request

REFERENCES:
- [Background] Ong SWX, Tan YK, Chia PY, Lee TH, Ng OT, Wong MSY, Marimuthu K. Air, Surface Environmental, and Personal Protective Equipment Contamination by Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) From a Symptomatic Patient. JAMA. 2020 Apr 28;323(16):1610-1612. doi: 10.1001/jama.2020.3227. PMID 32129805
- [Background] Hui DS, Chow BK, Lo T, Tsang OTY, Ko FW, Ng SS, Gin T, Chan MTV. Exhaled air dispersion during high-flow nasal cannula therapy versus CPAP via different masks. Eur Respir J. 2019 Apr 11;53(4):1802339. doi: 10.1183/13993003.02339-2018. Print 2019 Apr. PMID 30705129
- [Background] Leung CCH, Joynt GM, Gomersall CD, Wong WT, Lee A, Ling L, Chan PKS, Lui PCW, Tsoi PCY, Ling CM, Hui M. Comparison of high-flow nasal cannula versus oxygen face mask for environmental bacterial contamination in critically ill pneumonia patients: a randomized controlled crossover trial. J Hosp Infect. 2019 Jan;101(1):84-87. doi: 10.1016/j.jhin.2018.10.007. Epub 2018 Oct 15. PMID 30336170
- [Background] Hui DS, Chow BK, Chu L, Ng SS, Lee N, Gin T, Chan MT. Exhaled air dispersion during coughing with and without wearing a surgical or N95 mask. PLoS One. 2012;7(12):e50845. doi: 10.1371/journal.pone.0050845. Epub 2012 Dec 5. PMID 23239991
- [Background] Johnson DF, Druce JD, Birch C, Grayson ML. A quantitative assessment of the efficacy of surgical and N95 masks to filter influenza virus in patients with acute influenza infection. Clin Infect Dis. 2009 Jul 15;49(2):275-7. doi: 10.1086/600041. PMID 19522650
- [Derived] Li J, Jing G, Fink JB, Porszasz J, Moran EM, Kiourkas RD, McLaughlin R, Vines DL, Dhand R. Airborne Particulate Concentrations During and After Pulmonary Function Testing. Chest. 2021 Apr;159(4):1570-1574. doi: 10.1016/j.chest.2020.10.064. Epub 2020 Nov 1. No abstract available. PMID 33144080